CLINICAL TRIAL: NCT00064792
Title: Investigation of Simvastatin Therapy in Smith-Lemli-Opitz Syndrome
Brief Title: Simvastatin Therapy in Smith-Lemli-Opitz Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forbes Porter, M.D. (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Forbes Porter, M.D., Clinical Director, NICHD, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 030225; 03-CH-0225
Record Dates: First submitted 2003-07-11; First posted 2003-07-14 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: Cholesterol; SLOS; HMG-COA Reductase Inhibitor; Malformation Syndrome; Mental Retardation; Smith-Lemli-Opitz Syndrome
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome; Intellectual Disability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OraPlus (Placebo Comparator)
  Interventions: Drug: OraPlus
- Simvastatin Susp (Active Comparator)
  Interventions: Drug: Simvastatin Susp.

INTERVENTIONS:
Drug: Simvastatin Susp. — During the simvastatin phase of the trial, therapy will be initiated at 0.5 mg/kg/day for six weeks and then increased to 1.0 mg/kg/day if adverse side effects are minimal or absent.
  Arms: Simvastatin Susp
Drug: OraPlus — During this trial and for two months prior, patients will be maintained on 150 mg/kg/day of dietary cholesterol (150 mg/ml in OraPlus) for the duration of the trial
  Arms: OraPlus

SUMMARY:
This study will evaluate the safety and effectiveness of simvastatin in treating children with Smith-Lemli-Opitz syndrome (SLOS). Patients with this inherited disease are deficient in an enzyme that converts a substance called 7-dehydrocholesterol (7-DHC) to cholesterol. Cholesterol synthesis is impaired, causing birth defects and mental retardation. This study will examine whether simvastatin can increase the amount of the deficient enzyme, thereby lowering 7-DHC and increasing cholesterol. It will examine the safety of simvastatin in affected children and its effects on their behavioral problems.

Children between 4 and 18 years of age with mild to typical SLOS may be eligible for this study. Participants will be evaluated at the NIH Clinical Center in Bethesda, MD, and at the Kennedy Krieger Institute in Baltimore, MD, upon admission to the study and again at 6, 12, 20, and 26 months. The visits will last 3 to 4 days, and will include a medical history and physical examination, photographs to document medical findings, and other procedures detailed below. In addition, blood samples will be collected at 1, 3, 9, 14, 15, 17, and 23 months. Parents will complete several questionnaires during the study. Procedures include the following:

* Simvastatin and cholesterol supplementation therapy. Patients take cholesterol supplements (50 milligrams per kilogram per day) plus simvastatin (0.5 mg/kg/day for 6 weeks and then 1 mg/kg/day) for 12 months, and cholesterol supplements plus a placebo for 12 months.
* Blood draws to check liver, muscle, and kidney function, hormone levels, vitamin D levels, blood counts, cholesterol and 7-DHC levels, and lipoprotein levels. Some extra blood is drawn for research purposes.
* Urine collection. Urine is collected using a toilet hat. For children who are not toilet trained, urine is collected in a bag taped to the skin with an adhesive.
* Electroretinogram (ERG) to measure the function of the retina, the light-sensitive tissue at the back of the eye. ERG is done under sedation. After adapting the child's eyes to the dark, an electrode is taped to the child's forehead, the surface of one eye is numbed with eye drops, and a contact lens is placed on the eye. The child looks inside a globe that emits a series of light flashes. The contact lens senses electrical signals generated by the retina when the light flashes. After the ERG, the patient has a full eye exam, including pupil dilation and photographs of the eye.
* Lumbar puncture (spinal tap) to collect a sample of cerebral spinal fluid (CSF). This procedure, done while the patient is sedated for the ERG, shows whether simvastatin affects brain cholesterol and chemical levels. Under local anesthetic, a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle.
* CRH stimulation test to detect hormone-related problems in cholesterol synthesis. The patient is given CRH, a hormone involved in cholesterol synthesis, through a plastic tube placed in a vein. Blood samples are collected through the same catheter to measure levels of other hormones involved in cholesterol production.
* Electroencephalogram (EEG) to look at the electrical activity (brain waves) of the child's brain.
* Activity monitoring. An activity monitor, which looks like and is worn like a watch, is used to record the child's level of activity for a 48-hour period.
* Urine pregnancy test at every visit for female patients over age 10.
* Skin swab for sterol (solid alcohol, such as cholesterol) analysis. An alcohol pad is rubbed lightly against the child's arm or thigh to collect skin cells.
* Stool collection. A small stool sample is collected from the child's diaper or, for children who are toilet trained, from a toilet "hat" like that used to collect urine.

DETAILED DESCRIPTION:
Smith-Lemli-Opitz syndrome (SLOS, RSH, OMIM #270400) is an autosomal recessive, multiple malformation, mental retardation syndrome due to an inborn error of cholesterol biosynthesis. Specifically, these patients have a deficiency of 3 beta-hydroxysterol Delta 7-reductase activity due to mutation of the 3 beta-hydroxysterol delta 7-reductase gene (DHCR7). This enzymatic deficiency impairs the conversion of 7-dehydrocholesterol (7-DHC) to cholesterol in the last step of cholesterol biosynthesis via the Kandutch-Russel biosynthetic pathway. The clinical manifestations of SLOS are extremely variable and the phenotypic spectrum is broad. At the severe end of the spectrum SLOS is a lethal disorder with multiple major congenital anomalies, and in mild cases SLOS combines minor physical stigmata with behavioral and learning disabilities. Based on clinical studies, the incidence of SLOS is on the order of 1/10,000 to 1/60,000. Molecular studies have shown a carrier frequency of about 1% for the most common SLOS mutant allele in North American populations. Currently therapy is based on dietary cholesterol supplementation. Although clinical improvement has been noted, serum cholesterol levels are rarely normalized and elevated serum 7-DHC levels persist. Because elevated 7-DHC levels may have toxic effects, treatment of SLOS patients with an HMG-CoA reductase inhibitor has been proposed. Two small (two-patient) open trials of simvastatin therapy in SLOS have been reported. One of these trials showed improved clinical status, decreased 7-DHC levels and increased cholesterol levels. The second trial showed decreased 7-DHC levels; however, treatment had to be discontinued in one patient with preexisting liver disease. The goal of this clinical research protocol will be to test the clinical efficacy and safety of simvastatin therapy in mild to classical SLOS patients using a double blinded, crossover design.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients with biochemically proven SLOS will be considered for this study.

EXCLUSION CRITERIA:

Patients will be excluded if they cannot travel to the NIH because of their medical condition.

Age less than 4 and older than 18.

Weight less than 10 kg.

Developmental delay too severe to obtain adequate behavioral evaluation.

Severe behavioral problems that preclude proper physical and laboratory medicine evaluation.

SLOS severity score greater than 30.

No biochemical diagnosis of SLOS.

No molecular conformation of SLOS.

Residual fibroblasts enzymatic activity less than 10% of control value (cholesterol synthesis as a fraction of total sterol synthesis).

Dehydrocholesterol/cholesterol ratio greater than 1.0.

Renal insufficiency.

Contraindications for simvastatin use:

History of hypersensitivity to simvastatin or other "statins."

Acute liver disease.

Persistent elevations of serum transaminase levels or persistent elevations of CPK.

Concomitant therapy with tetralol-class calcium channel blockers (such as mibefradil).

Pregnancy or lactation.

History of rhabdomyolysis or myopathy.

Concomitant therapy with other drugs associated with myopathy (such as gemfibrozil or other fibrates, niacin) or metabolism by the P450 isoform 3A4 system (such as cyclosporin, itraconazole, ketoconazole, macrolide antibiotics, or nefazodone (Serzone)).

Warfarin-type anticoagulant therapy.

Severe cataracts.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2003-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Porter FD. RSH/Smith-Lemli-Opitz syndrome: a multiple congenital anomaly/mental retardation syndrome due to an inborn error of cholesterol biosynthesis. Mol Genet Metab. 2000 Sep-Oct;71(1-2):163-74. doi: 10.1006/mgme.2000.3069. PMID 11001807
- [Background] Kelley RI, Hennekam RC. The Smith-Lemli-Opitz syndrome. J Med Genet. 2000 May;37(5):321-35. doi: 10.1136/jmg.37.5.321. PMID 10807690
- [Background] Kelley RI. A new face for an old syndrome. Am J Med Genet. 1997 Jan 31;68(3):251-6. doi: 10.1002/(sici)1096-8628(19970131)68:33.0.co;2-p. No abstract available. PMID 9024554
- [Derived] Thurm A, Tierney E, Farmer C, Albert P, Joseph L, Swedo S, Bianconi S, Bukelis I, Wheeler C, Sarphare G, Lanham D, Wassif CA, Porter FD. Development, behavior, and biomarker characterization of Smith-Lemli-Opitz syndrome: an update. J Neurodev Disord. 2016 Apr 5;8:12. doi: 10.1186/s11689-016-9145-x. eCollection 2016. PMID 27053961
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-CH-0225.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 subjects were consented and enrolled. 18 of 23 completed both arms of the study.
Pre-assignment Details: Each arm of the trial (placebo then simvastatin or simvastatin then placebo) was 12 months in length. The wash out period between phases was 2 months. Each subject served as own control.
Groups:
- Placebo Followed by Simvastatin: Subjects maintained cholesterol intake of 150mg/kg/day for 12 months. After a 2 month wash out period, they then received Simvastatin 1mg/kg/day (after starting at 0.5mg/kg/day for 6 weeks) in addition to cholesterol.
- Simvastatin Followed by Placebo: Subjects first received Simvastatin (1mg/kg/day after starting at 0.5mg/kg/day for 6 weeks) in addition to cholesterol 150mg/kg/day for 12 months. After a 2 month wash out period, they then continued with cholesterol supplementation only.
Period: Overall Study
Arm/Group | Placebo Followed by Simvastatin | Simvastatin Followed by Placebo
Started | 13 | 10
Completed | 8 | 10
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Followed by Simvastatin: During the placebo phase, subjects were given a daily dose of an oral suspension not containing active drug. All subjects continued taking cholesterol suspension at 150mg/kg/day.
- Simvastatin Followed by Placebo: Subjects began this phase by taking 0.5mg/kg/day of an oral suspension with active drug for 6 weeks followed by a daily dose of 1mg/kg/day. Subjects continued taking 150mg/kg/day of cholesterol suspension.
- Total: Total of all reporting groups
Arm/Group | Placebo Followed by Simvastatin | Simvastatin Followed by Placebo | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 10 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.576388889 (4.464005643) | 7.775 (2.286247802) | 8.175694444 (3.58400024)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Serum Cholesterol to Total Sterol Ratio
Description: Total serum cholesterol (mg/dL) divided by the sum of all sterols (cholesterol plus its precursors, 7-dehydrocholesterol - 7DHC, and 8-dehydrocholesterol- 8DHC - in mg/dL).
Time Frame: 1 year after therapy.
Population: The number of participants was determined by the total number of participants to complete both phases of the trial (n=18).
Measure: Mean (Standard Deviation); unit: percent total cholesterol
Groups:
- Not Simvastatin: During the placebo phase, subjects were given a daily dose of an oral suspension (OraPlus) not containing active drug. All subjects continued taking cholesterol suspension at 150mg/kg/day.
- Simvastatin: Subjects began this phase by taking 0.5mg/kg/day of an oral suspension with active drug for 6 weeks followed by a daily dose of 1mg/kg/day. Subjects continued taking 150mg/kg/day of cholesterol suspension.
Arm/Group | Not Simvastatin | Simvastatin
Number analyzed (Participants) | 18 | 18
percent total cholesterol | 90.82 (8.52) | 93.99 (5.36)
Statistical Analysis 1: Comparison: Not Simvastatin vs Simvastatin; The primary outcome variable will be the serum cholesterol/total sterol ratio; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

2. Secondary Outcome: Cerebral Spinal Fluid Dehydrocholesterol to Total Sterol Ratio
Description: Percent of 7-dehydrocholesterol + 8-dehydrocholesterol as a fraction of the total sterols (cholesterol + 7-dehydrocholesterol + 8-dehydrocholesterol measured in cerebral spinal fluid
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percent of total sterols
Arm/Group | Not Simvastatin | Simvastatin
Number analyzed (Participants) | 18 | 18
percent of total sterols | 5.898 (4.684) | 5.154 (3.067)
Statistical Analysis 1: Comparison: Not Simvastatin vs Simvastatin; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: muscle pain, elevated CK
Groups:
- OraPlus: During the placebo phase, subjects were given a daily dose of an oral suspension not containing active drug. All subjects continued taking cholesterol suspension at 150mg/kg/day.
- Simvastatin Susp: Subjects began this phase by taking 0.5mg/kg/day of an oral suspension with active drug for 6 weeks followed by a daily dose of 1mg/kg/day. Subjects continued taking 150mg/kg/day of cholesterol suspension.
Arm/Group | OraPlus | Simvastatin Susp
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | OraPlus (N=23) | Simvastatin Susp (N=23)
Muscle Pain and Elevated CK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/10 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes